CLINICAL TRIAL: NCT01053806
Title: A PHASE 2, SINGLE ARM STUDY TO DETERMINE THE SAFETY AND EFFICACY OF AZACITIDINE, AND LENALIDOMIDE IN HIGHER RISK MYELODYSPLASTIC SYNDROME
Brief Title: Safety And Efficacy Of Azacitidine, and Lenalidomide In Higher Risk Myelodysplastic Syndrome
Acronym: ViLen 001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-10-MM-0437-09-CTIL
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Myelodysplastic Syndrome
Keywords: MDS; Lenalidomide; 5-Azacytidine.; ORR; PFS; myelodysplastic syndrome.High risk.
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; Lenalidomide

INTERVENTIONS:
Drug: 5-Azacytidine and Lenalidomide — Induction:5-Azacytidine 75mg/m2/d S.C.or I.V. days 1-5 every 28 days a cycle for 6 cycles and Lenalidomide 10mg/d orally days 6-28 every cycle for 6 cycles Consolidation: 5-Azacytidine 75mg/m2/d S.C.or I.V. days 1-5 every 28 days for 6 cycles Maintenance: Lenalidomide 10mg/d orally days 1-21 every cycle of 28 days for 13 cycles.

SUMMARY:
To evaluate the overall response rate of the combination of 5-azacitidine + Lenalidomide in high risk MDS patients (INT-2 and High risk defined by IPSS), and patients with low and int-1 who are considered to be at high risk due to unfavorable additional factors.

* To evaluate the safety of the combination of 5-azacitidine + Lenalidomide in high risk MDS patients.
* To evaluate the hematological improvement rate.
* To evaluate the cytogenetic response rate.
* To evaluate the Progression free survival (PFS).
* To assess Quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
2. Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
3. Patient is older than 18 years at the time of signing the informed consent.
4. Female subjects of childbearing potential† must:

   Understand that the study medication could have a potential teratogenic risk (Lenalidomide is structurally related to thalidomide which is a known human teratogenic active substance that causes severe life-threatening birth defects. Lenalidomide induced in monkeys malformations similar to those described with thalidomide)

   Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhoea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. The following are effective methods of contraception • Implant - Levonorgestrel-releasing intrauterine system (IUS)
   * Medroxyprogesterone acetate depot • Tubal sterilisation • Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses • Ovulation inhibitory progesterone-only pills (i.e., desogestrel)

   Combined oral contraceptive pills are not recommended. If a subject was using combined oral contraception, she must switch to one of the methods above. The increased risk of VTE continues for 4 to 6 weeks after stopping combined oral contraception.

   prophylactic antibiotics should be considered at the time of insertion particularly in patients with neutropenia due to risk of infection

   o Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mIU/ml not more than 3 days from the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.

   Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These tests should be performed not more than 3 days before the start of next treatment. This requirement also applies to women of childbearing potential who practice complete and continued abstinence

   Male subjects must Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.

   Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.

   All subjects must Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.

   Agree not to share study medication with another person and to return all unused study drug to the investigator
5. Patient was diagnosed with Myelodysplastic syndrome, INT-2 or HIGH risk according IPSS score, Low risk and INT-1 risk patients that meet all of the following criteria may also be included into the trial when they meet the following criteria:

   - Resistant to EPO

   - No transfusion independence achieved with lenalidomide treatment alone
   * RBC transfusion dependant
   * cytogenetic abnormalities: del 5q, chromosome 7, 5q with complex karyotypes
6. Bone marrow aspiration examination including cytogenetics performed up to 12 months before patient signing informed consent.
7. Patient was defined as erythropoietin resistant (not increasing Hb level after 8 weeks of erythropoietin treatment in the past or is not planed to receive erythropoietin in study period.)
8. Patient has a Performance status 0-2 (WHO).(see appendix V)
9. Patient has a life-expectancy > 6 months
10. Patient has negative serology for: active infectious hepatitis type B or C, or HIV infection.
11. Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1):

    * Platelet count ≥ 25 x 109/L without transfusion support within 7 days before the test.
    * Absolute neutrophil count (ANC) ≥ 0.5 x 109/L without the use of growth factors.
    * Aspartate transaminase (AST): ≤2.5 x the upper limit of normal (ULN).
    * Alanine transaminase (ALT): ≤ 2.5 x the ULN.
    * Total bilirubin: ≤ 1.5 x the ULN.
    * serum creatinine: ≤ 2 X the ULN

Exclusion Criteria:

1. Previous treatment with anti-MDS therapy in the last 2 months (including growth factors, does not include blood transfusions).
2. Any serious medical condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he or she participates in this study or confounds the experimental ability to interpret data from the study.
3. Pregnant or lactating females.
4. Prior history of malignancies, other than MDS, unless the subject has been free of the disease for ≥ 3 years. Exceptions include the following: Basal cell carcinoma of the skin, Squamous cell carcinoma of the skin, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histologic finding of prostate cancer (TNM stage of T1a or T1b)
5. Patients previously diagnosed as bearing deep venous thrombosis or arterial thromboembolic event within the latest 6 months, or bearing a clear contra indication for anti-platelet or anticoagulant therapy or bearing a high risk of bleeding complications are ineligible for the study protocol.
6. Bone marrow blast count > 30%
7. low risk MDS according IPSS with no additional features appearing in inclusion criteria number 5
8. Total bilirubin > 1.5 x ULN
9. AST/ALT > 2.5 x ULN
10. Serum creatinine > 2 x ULN
11. Known allergy or intolerance to Lenalidomide or 5-azacitatidine or any of the exipients
12. Use of chemotherapeutic drugs or biologic agents or steroids in the last 3 months.
13. Administration of investigational drugs in the last 3 month
14. Known neuropathy

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years

SECONDARY OUTCOMES:
PFS | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of internal medicine A, Tel Aviv, Israel